CLINICAL TRIAL: NCT02628262
Title: Fundus Autofluorescence Images in Gas-filled Eyes Immediately After Macular Hole Surgery
Brief Title: Fundus Autofluorescence After Macular Hole Surgery
Status: Completed | Type: Observational
Sponsor: Makoto Inoue (Other)
Responsible Party: Sponsor-Investigator, Makoto Inoue, Professor of Ophthalmology, Kyorin University
Organization: Kyorin University (Other)
Other Study IDs: Kyorineye020
Record Dates: First submitted 2015-12-06; First posted 2015-12-11 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Macular Hole
Keywords: Macular hole
MeSH Terms: conditions — Retinal Perforations | interventions — Vitrectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Vitrectomy with internal limiting membrane removal and gas tamponade — Vitrectomy with internal limiting membrane removal and gas tamponade

SUMMARY:
Funds autofluorescence (FAF) indicates hyper fluorescence at the macular hole in the patients with macular hole. Investigators investigate the association between FAF and visual acuity, recovery of foveal microstructure, and FAF in surgically closed macular holes.

DETAILED DESCRIPTION:
Ultrawide angle FAF images were taken in 27 eyes before and after macular hole surgery and compared with swept source optical coherence tomographic (SS-OCT) images.

ELIGIBILITY:
Inclusion Criteria:

* The patients were followed more than 6 months.

Exclusion Criteria:

* The patient were followed less than 6 months.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Optos ultrawide angle FAF images were taken in 27 eyes before and after MH surgery and compared with swept source optical coherence tomographic (SS-OCT) images.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2013-04; Primary Completion 2015-04 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Visual acuity before and after surgery | Changes from baseline to 1,3, 6 months
  Vision

SECONDARY OUTCOMES:
Fundus autofluorescence at the macula | Changes from baseline up to 6 months
  Fundus autofluorescence at the macula

CONTACTS AND LOCATIONS:
Locations (1):
- Makoto Inoue, Mitaka, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No